CLINICAL TRIAL: NCT03143010
Title: Comparison of Different Doses of Dexmedetomidine Effect in the Duration of Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Dexmedetomidine12
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Spinal Anesthesia Duration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Placebo Comparator): intrathecal Dexmedetomidine received 3mL (15mg) of 0.5% levobupivacaine +0.5mL normal saline .
  Interventions: Drug: intrathecal Dexmedetomidine
- 1.5 DEX (Experimental): Dexmedetomidine 1.5 micrograms received 3mL (15mg) of 0.5% levobupivacaine +0.5ml (1.5μg) dexmedetomidine
  Interventions: Drug: Dexmedetomidine 1.5 micrograms
- 3 DEX (Experimental): Dexmedetomidine 3 micrograms received 3mL (15mg) of 0.5% levobupivacaine +0.5ml (3μg) dexmedetomidine
  Interventions: Drug: Dexmedetomidine 3 micrograms
- 5 DEX (Experimental): Dexmedetomidine 5 micrograms received 3mL (15mg) of 0.5% levobupivacaine +0.5ml (5μg) dexmedetomidine
  Interventions: Drug: Dexmedetomidine 5 micrograms

INTERVENTIONS:
Drug: intrathecal Dexmedetomidine — injection of different doses of Dexmedetomidine intrathecally received 3mL (15mg) of 0.5% levobupivacaine +0.5mL normal saline.
  Other Names: saline intrathecally
  Arms: control group
Drug: Dexmedetomidine 1.5 micrograms — injection of different doses of Dexmedetomidine intrathecally in the form of 3mL (15mg) of 0.5% levobupivacaine +0.5mLof 1.5 micrograms of Dexmedetomidine.
  Other Names: Dexmedetomidine 1.5 micrograms intrathecally
  Arms: 1.5 DEX
Drug: Dexmedetomidine 3 micrograms — injection of different doses of Dexmedetomidine intrathecally in the form of 3mL (15mg) of 0.5% levobupivacaine +0.5mLof 3 micrograms of Dexmedetomidine.
  Other Names: Dexmedetomidine 3 micrograms intrathecally
  Arms: 3 DEX
Drug: Dexmedetomidine 5 micrograms — injection of different doses of Dexmedetomidine intrathecally in the form of 3mL (15mg) of 0.5% levobupivacaine +0.5mLof 5 micrograms of Dexmedetomidine.
  Other Names: Dexmedetomidine 5 micrograms intrathecally
  Arms: 5 DEX

SUMMARY:
Small doses of dexmedetomidine1.5,3, 5µg used in combination with bupivacaine, in humans for spinal anesthesia has been shown to produce a more rapid onset of motor block, and a longer duration of motor and sensory block with preserved hemodynamic stability and lack of sedation.

DETAILED DESCRIPTION:
Spinal anesthesia has many advantages such as reducing the metabolic stress response to surgery, reduction in blood loss, decrease in the incidence of venous thromboembolism, reduction in pulmonary compromise (particularly in patients with advanced pulmonary disease),return of bowel function rapidly, allow hospital discharge early and the ability to monitor the patient's mental status, but the limited duration of action is one of its disadvantages. Intrathecal α2-agonists prolong the duration of action of local anesthetics and reduce the total required dose.(1, 2) Dexmedetomidine is a centrally acting highly specific α2 -agonist and its α2/α1 selectivity are 8 times higher than that of clonidine.(3) It is commonly used as a sedative, preemptive analgesic,(4) to decrease the incidence of postoperative nausea, vomiting (PONV)(5) and to maintain stable hemodynamics(6). It also has been used as an additive to local anesthetics in peripheral nerve blocks, brachial plexus block7, subarachnoid anesthesia and caudal anesthesia (8).

Local anesthetics have been widely used in medical practice to produce anesthesia, analgesia and for pain management. Nowadays, minor surgical operations have been done under local anesthesia outside the operating theaters, in this area monitoring and resuscitation facilities of the case are suboptimal compared to operating rooms. The complications of local anesthesia are different from localized reactions such as urticaria, edema, and dermatitis to systemic absorption leading to severe cardiovascular collapse and neurological toxicity. The incidence of local anesthetics to produce systemic toxicity decreased in the past 30 years, from 0.2 to 0.01 %.( 9) Recently, patient safety changes a clinician's perspective on understanding the pharmacology of drug interactions and complications of local anesthetics. The safety of local anesthetic usage has improved owing to the introduction of newer agents (eg; Ropivacaine and Levobupivacaine). (10) Levobupivacaine is a long-acting local anesthetic similar to that of Bupivacaine in a pharmacological structure. Bupivacaine, a widely used local anesthetic in regional anesthesia presents in a commercial preparation as a racemic mixture (50:50) of its two enantiomers, Levobupivacaine, S (-) isomer and destroy- bupivacaine, R (+) isomer.

Levobupivacaine has been shown to have a safer pharmacological profile (11) with less cardiac and neurotoxic adverse effects. (12) Small doses of dexmedetomidine 5µg used in combination with Levobupivacaine, in humans for spinal anesthesia has been shown to produce a more rapid onset of motor block, and a longer duration of motor and sensory block with preserved hemodynamic stability and lack of sedation2.

ELIGIBILITY:
Inclusion Criteria:

* Patients' physical status by the American Association of Anesthesiology (ASA): ASA I, II, III, undergoing Lower abdominal surgeries of maximum duration 2hrs

Exclusion Criteria:

* patients who refuse regional anesthesia or patient with bleeding tendency, taking α2- adrenergic agonist, labile hypertension, uncontrolled cardiac disease, heart block/dysrhythmia, difficulty in communication e.g. mental retardation or deafness, body weight more than 120kg or height less than 150cm, allergic to any of the drugs used in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-07 (Actual); Primary Completion 2017-07-30 (Estimated); Study Completion 2017-07-30 (Estimated)

PRIMARY OUTCOMES:
duration of sensory block | 6 hours
  time from onset of spinal to full recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided